CLINICAL TRIAL: NCT00833859
Title: A Phase 2 Study of GTX-SRS: Neoadjuvant Gemcitabine, Docetaxel, and Capecitabine in Combination With Stereotactic Radiosurgery for Borderline Resectable Pancreatic Cancer
Brief Title: Neoadjuvant Gemcitabine, Docetaxel, and Capecitabine in Combination With Stereotactic Radiosurgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Abandoned - Lack of funding after only 2 patients enrolled
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15587; IST 14091 (Other: Sanofi-Aventis US Inc.)
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2011-05-26 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2013-12

CONDITIONS: Pancreatic Neoplasms
Keywords: stereotactic radiosurgery; borderline resectable pancreatic cancer; gastrointestinal; pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Docetaxel; Capecitabine; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy followed by Radiation Treatment (Experimental): GTX-SRS: Gemcitabine, Taxotere, Xeloda (GTX)-Stereotactic Radiosurgery (SRS)
  Interventions: Drug: GTX (gemcitabine, docetaxel and capecitabine); Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Drug: GTX (gemcitabine, docetaxel and capecitabine) — GTX: 21 day cycle x 2 Gemcitabine 750mg/m2 on days 4 and 11 Taxotere® (docetaxel) 30 mg/m2 on days 4 and 11 Xeloda® (capecitabine) 750 mg/m2 on days 1-14
  Other Names: Gemcitabine; Taxotere®; docetaxel; Xeloda®; capecitabine
Radiation: stereotactic body radiation therapy — stereotactic body radiation therapy (SBRT) 25
  Other Names: SBRT

SUMMARY:
The purpose of this study is to find out if a program of intensive chemotherapy with gemcitabine, docetaxel and capecitabine followed by an advanced form of focused radiation aimed at the patient's tumor followed by more chemotherapy can increase the chances that the patient's pancreatic tumor can be removed completely.

DETAILED DESCRIPTION:
* Cycle 1 and 2:

  * Days 4, 11 and 25, 32 ....gemcitabine 750 mg/m^2 intravenous piggy back (IVPB) over 30 min
  * Days 4, 11 and 25, 32 ....docetaxel 30 mg/m^2 IVPB over 1 hour
  * Days 1-14 and 22-35 ....capecitabine 750 mg/m^2 oral twice daily
  * Each cycle is 21 days long
* SRS: Day 43 ....25 Gy single fraction to the pancreatic tumor gross target volume
* Cycle 3 and 4:

  * Days 54, 61 and 75, 82 ....gemcitabine 750 mg/m^2 IVPB over 30 min
  * Days 54, 61 and 75, 82 ....docetaxel 30 mg/m^2 IVPB over 1 hour
  * Days 51-64 ....capecitabine 750 mg/m^2 oral twice daily
  * Each cycle is 21 days long
* Surgery: Exploratory laparotomy or laparoscopy followed by pancreaticoduodenectomy or central pancreatectomy with or without vein resection and reconstruction as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed pancreatic adenocarcinoma that is borderline resectable disease. Borderline resectable lesions are defined as:

  * circumferential tumor abutment with the superior mesenteric vein (SMV) or portal vein (PV) or SMV/PV confluence over < 180o.
  * circumferential tumor abutment with the superior mesenteric artery (SMA) over < 180o.
  * Short segment encasement (360o) of the PV or SMV that is amenable to partial vein resection and reconstruction.
  * encasement of the gastroduodenal artery up to the origin of the hepatic artery
* Patients must have measurable disease.
* No previous chemotherapy or radiation to the pancreas.
* Eastern Cooperative Oncology Group (ECOG) performance status <2 (Karnofsky >60%.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >3,000/μL
  * absolute neutrophil count >1,000/μL
  * platelets >100,000/μL
  * creatinine within normal institutional limits - OR - creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
  * total bilirubin < institutional upper limit of normal (ULN). Patients may have biliary stents or drains to lower total bilirubin to this range.
  * Aspartate Aminotransferase (AST) serum glutamic oxaloacetic transaminase(SGOT) / alanine aminotransferase (ALT) serum glutamic pyruvic transaminase(SGPT) AST and ALT may be up to 2.5 times ULN if alkaline phosphatase < ULN; or alkaline phosphatase may be up to 4 times ULN if AST and ALT are < ULN.
* Has a negative serum or urine pregnancy test within 7 days prior to initiation of therapy (female patients of childbearing potential). Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Patients will agree to continue contraception for 30 days from the date of the last study drug administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with metastatic disease are ineligible. Patients who have had prior chemotherapy for pancreatic adenocarcinoma.
* Patients who have received prior radiation to an abdominal site are not eligible.
* Prior malignancy in the last 3 years, except basal cell carcinoma, squamous cell or in-situ cervical cancer.
* Patients with peripheral neuropathy > grade 2.
* Patients with a history of severe hypersensitivity reaction to Taxotere (docetaxel), other drugs formulated with polysorbate 80, gemcitabine, or capecitabine.
* Patients may not be receiving any other investigational agents.
* ECOG PS 3-4
* Pregnant women are excluded from this study because gemcitabine, capecitabine, and docetaxel are Class D agents with the potential for teratogenic or abortifacient effects.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* creatinine clearance < 30 ml/min (Cockcroft-Gault method).
* Patients must not have any comorbid inflammatory conditions of the bowel such as Crohn's Disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Springett, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy Followed by Radiation Treatment: Gemcitabine, Taxotere, Xeloda (GTX)-Stereotactic Radiosurgery (SRS). GTX: 21 day cycle x 2 Gemcitabine 750mg/m2 on days 4 and 11 Taxotere® (docetaxel) 30 mg/m2 on days 4 and 11 Xeloda® (capecitabine) 750 mg/m2 on days 1-14. Stereotactic body radiation therapy (SBRT) 25.
Period: Overall Study
Arm/Group | Chemotherapy Followed by Radiation Treatment
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy Followed by Radiation Treatment
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Resectability
Description: The intent was to have 33 Evaluable Participants and measure the number of surgical resections with negative margins, ie. R0 resection rate. The new treatment would be of interest if the resectability rate was at least 30%. R0 resections were to be scored as those resections in which the common bile duct margin, pancreatic resection margin, retroperitoneal margin were negative for tumor involvement.
Time Frame: 6 months per patient
Population: Data for this study was not collected because the study was abandoned after two enrollments due to funding being cancelled.
Arm/Group | Chemotherapy Followed by Radiation Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs).
Description: Investigators planned to review the occurrences of AEs and SAEs according severity by NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0, Acute GI toxicity by Radiation Therapy Oncology Group (RTOG) Gastrointestinal (GI) toxicity scale.
Time Frame: 6 months per patient
Population: as for outcome 1
Arm/Group | Chemotherapy Followed by Radiation Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Objective Response
Description: Investigators planned to prospectively evaluate the ability of serum CA19-9 response and positron-emission tomography (PET) / computed tomography(CT) response to predict pathologic treatment response to GTX-SBRT and to determine the correlation of standardized uptake value (SUV) uptake on PET to fiducial marker placement.
Time Frame: 6 months per patient
Population: as for outcome 1
Arm/Group | Chemotherapy Followed by Radiation Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Overall Survival
Description: We intended to track the number of participants with overall survival at the projected end of the study period. The study was terminated prematurely.
Time Frame: 6 months per patient
Population: as for outcome 1
Arm/Group | Chemotherapy Followed by Radiation Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Chemotherapy Followed by Radiation Treatment
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy Followed by Radiation Treatment (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (5) — 1 of 5 events probably related, 4 definitely related
Intermittent hypotension (Cardiac disorders) | 1 (1) — Unrelated
Pale skin (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Itchy rash (Skin and subcutaneous tissue disorders) | 1 (1) — Related
Hand foot syndrome (Skin and subcutaneous tissue disorders) | 2 (3) — Related
Anorexia (Gastrointestinal disorders) | 1 (2) — Unrelated
Constipation (Gastrointestinal disorders) | 1 (2) — Unrelated
Nausea (Gastrointestinal disorders) | 1 (1) — Unrelated
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Dizziness/lightheadedness (General disorders) | 1 (1) — Unrelated
Presyncope (General disorders) | 1 (1) — Unrelated
Chest tightness (General disorders) | 1 (1) — Unrelated
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (3) — Unrelated
Anemia (Blood and lymphatic system disorders) | 1 (1) — Related
Increased fatigue (General disorders) | 1 (1) — Related
Insomia (General disorders) | 1 (1) — Unrelated
Cracks on lips (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Cracks on feet (Skin and subcutaneous tissue disorders) | 1 (1) — Possibly related
Red peeling spots on arms (Skin and subcutaneous tissue disorders) | 1 (1) — Related
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) — Related
Dehydration (Gastrointestinal disorders) | 1 (2) — Unrelated
Yellow stools (Gastrointestinal disorders) | 1 (1) — Unrelated
Hemorrhoid (Gastrointestinal disorders) | 1 (1) — Unrelated
Malabsorption (Gastrointestinal disorders) | 1 (1) — Unrelated
Mouth sores (Gastrointestinal disorders) | 1 (1) — Related
Intermittent nausea (Gastrointestinal disorders) | 1 (1) — Unlikely that it is related
Taste alteration (Gastrointestinal disorders) | 1 (1) — Related
Calf tightness (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Sort throat/redness (General disorders) | 1 (1) — Related
Voice changes (raspy) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Possibly related

LIMITATIONS AND CAVEATS:
Early termination of study due to termination of funding. The study was closed to accrual on 12/17/09 and final closed on 3/12/10. The sample size goal of 33 evaluable participants could not be met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No